CLINICAL TRIAL: NCT02045459
Title: Assessment of Perfusion Reserve and Effects of Exercise in Microvascular Angina
Brief Title: Microvascular Disease Exercise Trial
Acronym: MOVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Astellas Pharma Global Development, Inc. (Industry); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jamieson Bourque, MD, Assistant Professor, Cardiovascular Medicine, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 16821; 1K23HL119620-01 (NIH)
Record Dates: First submitted 2014-01-17; First posted 2014-01-24 (Estimated); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Coronary Microvascular Disease
Keywords: Microvascular Disease; Exercise; Angina; Chest pain
MeSH Terms: conditions — Microvascular Angina; Motor Activity; Angina Pectoris; Chest Pain | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exercise Program and Medical Therapy (Experimental): All subjects randomized to this arm will be given intensive medical therapy including - Isosorbide mononitrate, Lisinopril, Carvedilol, and Simvastatin. After 8 weeks of ONLY medication therapy, the subjects will begin a intensive exercise program. This will be supervised on site at UVA. Also, on days that the subject is not being supervised, they will be required to keep a journal of their exercise at home.
  Interventions: Behavioral: Exercise Program

INTERVENTIONS:
Behavioral: Exercise Program — Subject will be exercising on a treadmill 3x/week. Subjects progress will dictate increases/decreases in time of exercise and pace.

SUMMARY:
For part of this study, we are collecting information from patients that have been experiencing the symptoms mentioned above. We are taking this information and creating a chest pain registry to follow trends and compare different patients having similar symptoms. We hope to gain insight into the quality of life, symptoms, and cardiac events of those who are having similar symptoms. The type of information we will collect includes: demographics, quality of life, levels of anxiety related to angina pain and cardiac events occurring within a 2 year period of time.

In addition, we are performing a cardiac stress MRI for research purposes to look at the blood flow in the small vessels in your heart. During the stress cardiac MRI, we will give you a medication called Regadenoson (Lexiscan) which "stresses" your heart by dilating the blood vessels to your heart. This drug is approved by the U.S. Food and Drug Administration (FDA) for this purpose. We will then be able to measure the myocardial perfusion reserve (MPR) which is a measure of blood flow through the small blood vessels to see if an abnormal MPR and small blood vessel disease is associated with an increased risk of cardiovascular events, such as heart attack. At this point, there is no specific therapy for small vessel disease. In addition we have phase II of this study which is to determine if exercise and intensive medical therapy together compared to intensive medical therapy alone improves pain from the heart and improves overall quality of life.

DETAILED DESCRIPTION:
Cardiac angina is a major source of morbidity, affecting more than 5% of the U.S. population.2 It leads to more than 1.5 million hospitalizations and $190 billion in costs yearly.3 Obstructive coronary artery disease (CAD) is the most common cause of angina. However, no obstructive CAD is found on elective coronary angiography in more than 50% of cases.4, 5 These patients with angina but no obstructive CAD are a heterogeneous group. Some have noncardiac explanations for their angina or nonobstructive epicardial abnormalities such as coronary spasm. However, many patients with angina and no obstructive CAD have microvascular dysfunction from endothelial dysfunction or microvascular obstructive disease as the cause. These patients have microvascular angina.

The coronary microvasculature is responsible for more than 70% of coronary resistance and thus plays a key role in regulating blood flow to match demand.6 Microvascular dysfunction can occur in the setting of dilated, hypertrophic, and restrictive cardiomyopathies. However, it is commonly seen in the setting of atherosclerotic risk factors or can be idiopathic.6, 7 Microvascular dysfunction is manifest as insufficient stress myocardial blood flow and/or reduced myocardial perfusion reserve (MPR), the ratio of stress flow to rest flow, in response to a stress such as vasodilator administration. Absolute myocardial blood flow and MPR can be assessed noninvasively with high precision and accuracy by cardiac magnetic resonance (CMR) imaging Reduced MPR in patients with angina is associated with significant morbidity, including a high risk of cardiac events, high medical costs, and a decreased quality of life.Despite the poor prognosis of this population, therapeutic options to reduce angina and improve MPR have not been well studied. Preliminary analysis shows that statins may improve endothelial function. ACE-inhibitors and beta-blockers improve symptoms in Syndrome X, a related disorder in which patients have angina, no obstructive CAD, and ischemic changes but a better prognosis. Therapeutic exercise has also been used in the Syndrome X population, improving exercise tolerance and endothelial function and reducing symptom severity.Improvements in MPR could be expected with exercise due to the reduced resting flow and increased MPR seen in healthy volunteers and improved endothelial function from increased nitric oxide bioactivity in patients with probable microvascular dysfunction. However, no studies have examined the effect of these medications or their synergism with exercise on MPR, aerobic capacity, anginal symptoms, or quality of life in patients with angina and reduced MPR. Identification of an effective therapy that improved symptoms and prognosis would have dramatic impact on this highly prevalent patient population.

The primary goal of this study is to characterize which patients with angina but no obstructive CAD have reduced MPR and test the effectiveness of intensive medical therapy plus a 12-week supervised exercise program versus intensive medical therapy alone to improve MPR, aerobic capacity, and the patient-centered outcomes of cardiac events, angina severity, and quality of life in this population with microvascular angina.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 85
* Anginal symptoms of chest pain, dyspnea on exertion, or other anginal equivalent suspected to be secondary to myocardial ischemia
* Coronary angiogram without obstructive epicardial coronary artery disease (≥50% epicardial stenosis or fractional flow reserve of <0.80) within 6 months prior to enrollment or date of CMR #1, whichever is later and without intervening signs or symptoms suggestive of new obstructive epicardial CAD.

Exclusion Criteria:

* Prior CABG (due to limitations of CMR quantitative perfusion in this population)
* Prior myocardial infarction (due to its effects on myocardial flow reserve)
* Hypertrophic or restrictive cardiomyopathy
* Coronary vasospasm
* Acute coronary syndrome unless concurrent coronary angiography reveals no epicardial stenoses of >50%
* Contraindications to CMR including - intracranial aneurysm clips, implantable pacemaker or defibrillator, metal cochlear/intraocular implants, any metallic implant not listed as magnetic resonance compatible, severe claustrophobia or other inability to tolerate a 30 minute CMR study
* GFR < 45 ml/min/1.73² (to avoid nephrogenic systemic fibrosis and iodinated contrast dye - mediated ATN) based on creatinine within 30 days of CMR #1
* Acute kidney injury, defined by the KDIGO Clinical Practice Guidelines as an increase in serum creatinine of ≥0.3 mg/dL within 48 hours, an increase in serum creatinine ≥1.5 times baseline thought to have occurred in the past 7 days, or a urine volume <0.5mL/kg/h for 6 hours
* Severe liver disease, paraproteinemia syndromes (such as multiple myeloma), hepatorenal syndrome, or planned liver transplantation (gadolinium contraindication)
* Pregnancy (assessed by serum beta- HCG prior to CMR) due to unclear gadolinium fetal effects
* Known hypersensitivity to regadenoson, or gadolinium
* Other contraindications to regadenoson (heart rate < 40 bpm, 2nd or 3rd degree heart block, sick sinus syndrome without a pacemaker, severe asthma or COPD with ongoing wheezing or hospitalization within the past 6 months, systolic blood pressure <90mmHg, recent use of dipyridamole, methylxanthine (such as aminophylline) or dipyridamole use within the past 48 hours, or caffeine within 12 hours)
* Atrial fibrillation with rapid ventricular response, frequent ectopy, or other contraindications to ECG gating
* Inability to provide informed consent
* Life expectancy of < 2 years

  3. List any restrictions on use of other drugs or treatments.
* Subject will be asked to refrain from use of caffeine for 12 hours and methylxanthines and dipyridamole for 48 hours prior to any administration of regadenoson. Subject may not participate if pregnant or breastfeeding.

Phase 2:

1. List the criteria for inclusion

   * Enrollment in phase #1.
   * MPR <2.0 ml/g/min on CMR #1.
2. List the criteria for exclusion

   •Unable to exercise.
3. List any restrictions on use of other drugs or treatments. Subject will be asked to refrain from use of caffeine for 12 hours and methylxanthines and dipyridamole for 48 hours prior to any administration of regadenoson. Subject may not participate if pregnant or breastfeeding.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2014-05; Primary Completion 2020-01-21 (Actual); Study Completion 2021-05-17 (Actual)

PRIMARY OUTCOMES:
Change in MPR on CMR imaging from baseline with intensive medical therapy + supervised exercise versus intensive medical therapy alone. | 20 weeks from first visit after consent is signed
  Determined with the use of a stress MRI after subject has been randomized and completed said randomized arm.

SECONDARY OUTCOMES:
Incremental change in MPR with exercise over intensive medical therapy alone in the exercise subgroup | 20 weeks after randomization
  Determined by the use of stress MRI after subjects have completed their arm of randomization
Identification of reduced MPR (<2.0 ml/g/min) and borderline reduced MPR | Within 30 days of screening visit
  This number is established by the use of a stress MRI

CONTACTS AND LOCATIONS:
Overall Officials: Jamieson Bourque, BA,MD,MHS, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States